CLINICAL TRIAL: NCT06571682
Title: Comparison of the Effect of Anesthesia Applied by Target Controlled Infusion Method and Inhalation Anesthesia Method on Patient Outcomes in Pediatric Patients Undergoing Laparoscopic Surgery
Brief Title: Comparison of Target Controlled Infusion Anesthesia and Inhalation Anesthesia in Pediatric Laparoscopic Surgeries
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem ÖZ GERGİN, Principal Investigator, TC Erciyes University
Other Study IDs: 2022/354
Record Dates: First submitted 2024-06-03; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Laparoscopic Surgery; Target Controlled Infusion
Keywords: Pediatric Laparoscopic Surgery; Target Controlled Infusion; Propofol; Sevoflurane
MeSH Terms: interventions — Anesthetics, Inhalation; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Intravenous Anesthesia Group: Patients will undergo anesthesia induction as routine after premedication. Once the target BIS level is reached (40-60) and muscle relaxation is achieved, the airway will be secured with an appropriately sized endotracheal tube or laryngeal mask (LMA).
  The effect zone target concentration of propofol will be adjusted to 3 mcg/ml with the HKI device.
  Patients will receive controlled ventilation with 50% oxygen/air, and mechanical ventilation parameters will be adjusted so that the end tidal carbon dioxide level (EtCO2) is 35-45 mmHg.
  Interventions: Device: Target Controlled Infusion
- Inhalation Anesthesia Group: Patients will undergo anesthesia induction as routine after premedication. The level of sevoflurane, an inhalation gas, will be adjusted so that BIS values are between 40-60. Patients will receive controlled ventilation with 50% oxygen/air, and mechanical ventilation parameters will be adjusted so that the end tidal carbon dioxide level (EtCO2) is 35-45 mmHg.
  Interventions: Drug: Inhalation anesthetic

INTERVENTIONS:
Device: Target Controlled Infusion — TCI (Target Controlled Infusion) is a method used to maintain the dose and rate of anesthesia drugs within a target concentration range set by the anesthetist. This system delivers drugs intravenously to the patient using a computer-controlled pump. The anesthetist adjusts the drug concentration to achieve the desired depth of anesthesia. This method provides more precise control over anesthesia and facilitates maintaining the depth of anesthesia within the desired range.
  Other Names: TCI
  Groups: Total Intravenous Anesthesia Group
Drug: Inhalation anesthetic — In the inhalation anesthesia group, maintenance sevoflurane anesthesia will be applied after routine induction.
  Other Names: Sevoflurane
  Groups: Inhalation Anesthesia Group

SUMMARY:
Comparison of Target Controlled Infusion Anesthesia and Inhalation Anesthesia in Pediatric Laparoscopic Surgeries

DETAILED DESCRIPTION:
In pediatric age group patients undergoing laparoscopic surgery, total intravenous anesthesia (TIVA) and inhalation anesthesia methods are used as anesthesia methods in the intraoperative period; It is compared in terms of its effects on blood pressure, pulse, postoperative awakening time and awakening agitation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 years
* Patients weighing over 10 kilograms
* Patients who will undergo inguinal hernia surgery
* ASA (American Society of Anesthesiologists) classification I and II pediatric patients.

Exclusion Criteria:

* Absence of systemic illness.
* ASA (American Society of Anesthesiologists) classification III and above pediatric patients.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3-12 with ASA I-II undergoing laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Modified Aldrete Scoring System | Aftet surgery 1 hour
  The effects on recovery were monitored within the first hour of the postoperative period using the Modified Aldrete Scoring System (MASS). Totally 0-10 points can be given by MASS. Higher scores predicts better recovery.

SECONDARY OUTCOMES:
Blood pressure (mmHg) | After surger 1 hour
  The blood pressure of the patients will be measured and recorded in mmHg at five-minute intervals from the beginning until the first postoperative hour.
Heart rate (beats/minute) | After surgey 1 hour
  The heart rate of the patients will be measured and recorded in mmHg at five-minute intervals from the beginning until the first postoperative hour.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem OZ GERGİN, MD, Study Director — TC Erciyes University